CLINICAL TRIAL: NCT06675474
Title: Saliva Versus All-Site Microbiome and Proteome Mapping in Periodontitis
Brief Title: Microbiome and Proteome Mapping in Periodontitis
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assoc. Prof., Aydin Adnan Menderes University
Other Study IDs: All-Site Mapping
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva, serum, gingival crevicular fluid and subgingival plaque
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Periodontitis: These patients had at least two interdental sites (at two non-adjacent teeth) with interproximal CAL ≥5 mm, along with PD ≥6 mm and RBL extending to the mid-third of the root or beyond. CAL was not originated from endodontic lesions draining through the marginal periodontium, dental caries extending into the cervical areas of the teeth, trauma-related gingival recession or distal bone loss in 2nd molars owing to extractions of 3rd molars. They had ≤4 teeth lost due to periodontitis.
  Interventions: Other: Clinical periodontal measurements; Other: Saliva sampling; Other: Serum Sampling; Other: GCF sampling; Other: Subgingival plaque sampling

INTERVENTIONS:
Other: Clinical periodontal measurements — Clinical periodontal measurements included PD, CAL, BOP (+/-), GI, and PI. Clinical recordings were performed at six points (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) of all teeth, except the 3rd molars.
Other: Saliva sampling — The whole unstimulated saliva samples were collected. Each participant was asked first to rinse the mouth completely with tap water for 2 minutes, wait for 10 minutes. Then the participants were requested to let the saliva pool in their floor of the mouth and to allow the saliva to drain passively into a falcon tube, 5 minutes.
Other: Serum Sampling — 5 ml of venous blood were taken from the antecubital vein by a standard venipuncture method.
Other: GCF sampling — GCF was collected from the six sites (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) per tooth, except the 3rd molars, via steril paper strips.
Other: Subgingival plaque sampling — Subgingival plaque was collected by inserting two standardized paper points (no:30) at six sites (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) per tooth, except the 3rd molars.

SUMMARY:
This study aimed to compare the microbiome and proteome profiles of saliva, serum and all periodontal sites in patients with periodontitis. Saliva, serum, gingival crevicular fluid and subgingival plaque were obtained from three patients with stage III, grade C periodontitis. Quantitative proteomics were performed for proteome analysis of saliva, serum and gingival crevicular fluid, whereas shotgun whole genome sequencing was performed for microbiome analysis in saliva, serum and plaque.

DETAILED DESCRIPTION:
Study Population: According to the 2017 World Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions, 3 systemically healthy and non-smoking patients with stage III, grade C periodontitis were included in this study. Clinical periodontal measurements included probing depth (PD), clinical attachment loss (CAL), the dichotomous scoring of bleeding on probing (BOP +/-), gingival index (GI), and plaque index (PI). All clinical parameters were recorded at six points (mesiobuccal, buccal, distobuccal, mesiopalatal palatal, and distopalatal) per tooth, except the 3rd molars, by a single investigator (B.A) using a manual periodontal probe. The percentage of radiographic bone loss (RBL) at the interproximal sites were calculated on the digital panoramic radiographs as the ratio of the distance between bone level and the cemento-enamel junction to the length of the root.

Sampling: Saliva, serum, gingival crevicular fluid (GCF) and subgingival plaque samples were collected 1 day following the clinical periodontal recordings. All samples were obtained in the morning between 8:30 am-10:30 am.

Firstly, the whole unstimulated saliva samples were collected. The participants were requested to refrain from eating, drinking (except water), chewing gum, brushing and flossing 2 hours before saliva collection. Then they were asked to let the saliva pool in their floor of the mouth and to allow the saliva to drain passively into a falcon tube, 5 minutes which was then stored directly at -80°C. On the day of analysis, 1 mL of thawed saliva was centrifuged at 4000 rpm at 4°C for 20 minutes.

To obtain serum samples, 5 ml of venous blood were taken from the antecubital vein by a standard venipuncture method. Serum was isolated by centrifugation at 1,500 g for 15 minutes at 4°C and then immediately frozen and stored at -80°C.

GCF was collected from the six sites (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) per tooth, except the 3rd molars, via steril paper strips. A paper strip was placed inside the pocket till a slight resistance was encountered and was left there for 30 seconds. The absorbed fluid volume was measured with a calibrated electronic instrument. Six GCF strips from each tooth were placed directly into an empty Eppendorf tube and stored at -80°C until analysis. On the day of analysis, strips resuspended in 480 μL PBS in an Eppendorf tube. The sample was shaken overnight at 600 rpm at 4°C, then centrifuged for 60 minutes at 4000 rpm at 4°C.

Subgingival plaque was collected by inserting two standardized paper points (no:30) at six sites (mesiobuccal, buccal, distobuccal, mesiopalatal, palatal, and distopalatal) per tooth, except the 3rd molars. Two paper points were placed into the pocket and left place for 10 seconds. Paper points from each tooth per quadrant were placed directly into an empty Falcon tube and stored at -80°C until analysis. On the day of analysis, each plaque sample was obtained by pooling material from multiple teeth and resuspending it in 50 μL PBS per strip in a Falcon tube. The sample was shaken overnight at 600 rpm at 4°C, then vortexed for 1 minute on a benchtop vortexer, and sonicated for 1 min. It was then centrifuged for 60 min. at 4000 rpm at 4°C. 1 mL of the supernatant was collected for an additional centrifuge step at 16,100 x g for 10 minutes at 4°C before pellets were collected for further analysis.

DNA Extraction and Quantification: DNA was extracted from 1 mL of saliva, paper point extracts, and serum using the GenElute bacterial genomic DNA kit as per established protocols. Sample concentrations were quantified using a Qubit 4 fluorometer and the Qubit™ dsDNA HS Assay Kit.

Library Preparation and Sequencing: DNA libraries were prepared for next generation sequencing according to the established protocols. Sequencing was performed on an Illumina NovaSeq 6000 platform 2x150b.

Bioinformatics Analysis for Microbiota: This procedure included assessments of alpha diversity, beta diversity, and LDA effect size in the taxonomic analysis.

Proteomics analysis: Quantitative proteomics were done according to the established protocols. Peptides were separated using a Thermo Scientific EASY-nLC 1200 system with a 15 cm, 75 µm-diameter silica emitter packed with ReproSil-Pur C18-AQ resin. Protein identification was performed using Scaffold v4.0. MS data were searched with Mascot against a customized database, which included the Homo sapiens Uniprot database, a 260-sequence MS contaminants database, and reversed sequences as a decoy. Search results were imported into Scaffold for validation, with filters set at 3.0% protein false discovery rate with a minimum of 2 peptides, and a 1.0% peptide false discovery rate.

Functional Analysis of Regulated Proteins & Statistical Analysis: We conducted enrichment analysis using the R software and the clusterProfiler package. Gene Ontology terms were identified from the 'Biological Process' database and ranked by statistical significance using hypergeometric distribution. Benjamini-Hochberg correction was applied, with significance thresholds set at p-value < 0.01 and q-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* No history of smoking
* At least 24 natural teeth (excluding 3rd molars)

Exclusion Criteria:

* Being diagnosed with diabetes mellitus, rheumatoid arthritis, cardiovascular system diseases, endocrine, immunologic, and mucocutaneous disorders
* Use of antibiotics, antihypertensives immunosuppressive, anti-inflammatory drugs and topical antiseptic solutions within the past 6 months
* Having periodontal treatment in the previous year
* Wearing removable partial dentures or orthodontic appliances
* Pregnant or nursing women

Ages: 43 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of three systemically healthy and non-smoking patients with stage III, grade C peridontitis (3 males; age range 43 to 60 years) were consecutively enrolled from the population seeking periodontal treatment for the first time at the Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University, Aydın, Turkey, between December 2019 to February 2020.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Host proteomics profiles from saliva, serum and GCF | 24 hours after clinical periodontal measurements
  Concentrations
Microbial profiles from subgingival plaque and saliva | 24 hours after clinical periodontal measurements
  Linear discriminant analysis scores

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan Bostanci, Principal Investigator — Karolinska Institutet
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)